CLINICAL TRIAL: NCT04930237
Title: RELISTOR's Effects on Opioid-Induced Constipation in Postoperative 1-2 Level Anterior Lumbar Interbody Fusion Patients: A Case-Control Study
Brief Title: RELISTOR's Effects on Opioid-Induced Constipation
Status: Withdrawn | Type: Observational
Why Stopped: PI request to close study
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 013.MBSI.2021.D
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: OIC
MeSH Terms: interventions — Dioctyl Sulfosuccinic Acid; Bisacodyl; Magnesium Hydroxide; magnesium citrate; Sennosides; Enema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Patients who receive RELISTOR
  Interventions: Drug: Relistor Injectable Product
- Observational Group: Patients that receive standard of care
  Interventions: Drug: Docusate Calcium; Drug: Bisacodyl; Drug: Milk of magnesia; Drug: Magnesium citrate; Drug: Senna; Drug: Enema

INTERVENTIONS:
Drug: Relistor Injectable Product — 12-mg RELISTOR to be administered as once-daily subcutaneous injections for 4 to 7 days
  Groups: Experimental Group
Drug: Docusate Calcium — Standard of care
  Groups: Observational Group
Drug: Bisacodyl — Standard of Care
  Groups: Observational Group
Drug: Milk of magnesia — Standard of Care
  Groups: Observational Group
Drug: Magnesium citrate — Standard of Care
  Groups: Observational Group
Drug: Senna — Standard of Care
  Groups: Observational Group
Drug: Enema — Standard of Care
  Groups: Observational Group

SUMMARY:
This will be a prospective case-control study of 40 patients undergoing 1-2 level ALIF procedures at Methodist Dallas Medical Center (MDMC). Patient records will be reviewed to identify details including demographics, comorbidities, procedure details, and the primary and secondary outcome metrics.

DETAILED DESCRIPTION:
RELISTOR is a legally marketed device and will be used off-label under the authority of a health care practitioner within a legitimate practitioner-patient relationship with the intent of the "practice of medicine".

The use of RELISTOR in the experimental group of this study meets all of the following conditions:

* is not intended to be reported to the FDA in support of a new indication for use or to support any other significant change in the labeling for the drug;
* it is not intended to support a significant change in the advertising for the product;
* it does not involve a route of administration or dosage level, use in a subject population, or other factor that significantly increases the risks (or decreases the acceptability of the risks) associated with the use of the drug product;
* it is conducted in compliance with the requirements for IRB review and informed consent [21 CFR parts 56 and 50, respectively];
* it is conducted in compliance with the requirements concerning the promotion and sale of drugs [21 CFR 312.7]; and
* it does not intend to invoke 21 CFR 50.24

Screening and Enrollment:

Patients will undergo two levels of screening: the initial screening and a post-operative OIC screening. The initial screening will involve all 1-2 level ALIF patients in the experimental group and observational group who will be approached to participate in the study before surgery. After eligible patients agree to participate and sign the ICF, all patients will then be asked to complete the PAC-SYM instrument about their constipation symptoms over the past 2 weeks.

Patients in both groups will undergo their 1-2 level ALIF procedure and then will undergo the post-operative OIC screen/rescreen (as needed) daily for acute OIC for a maximum of 3 days (i.e., postoperative days 2 - 4). Patients who are found to have acute OIC will be designated to the experimental and observational treatment regimens accordingly to Study Treatment Regimens.

If a patient does not have acute OIC after they are rescreened on postoperative day 4, are discharged, or do not meet the inclusion criteria, will be placed in the not-constipated or post-operative screen failure group.

ELIGIBILITY:
Inclusion Criteria:

Experimental Group (initial screen):

* Age 18 years or older
* Inpatient who will undergo a 1-2 level ALIF procedure with Dr. Richard Meyrat
* Are not pregnant or lactating
* Does not have a history of drug abuse within the past 2 years
* Does not have a gastrointestinal ostomy

Experimental Group (post-operative OIC screen/rescreen)

* Actively constipated (i.e., no BM in last 48 hours, difficult having a spontaneous BM, or inability to have a spontaneous BM)
* Receiving mu-agonist opioids
* Expected to require daily opioid analgesics for at least 7 days following enrollment
* Have not received or discontinued use of any laxatives, enemas and/or promotility agents within 48 hours of enrollment and the first dose of RELISTOR. Stool softeners are permitted.
* Does not have a known hypersensitivity to methylnaltrexone, naltrexone, or naloxone

Observational Group (initial screen):

* Age 18 years or older
* Inpatient who will undergo 1-2 level ALIF procedure with Dr. Graham
* Are not pregnant or lactating
* Does not have a history of drug abuse within the past 2 years
* Does not have a gastrointestinal ostomy

Observational Group (post-operative OIC screen/rescreen):

* Actively constipated (i.e. no BM in last 48 hours, difficulty having a spontaneous BM, or inability to have a spontaneous BM)
* Receiving mu-agonist opioids
* Expected to require daily opioid analgesics for at least 7 days following enrollment

Exclusion Criteria:

Experimental Group (post-operative OIC screen/rescreen):

Exclude patients with:

* Fecal impaction
* Mechanical bowel obstruction
* Constipation not attributed to post-procedural opioid use
* Calculated creatinine clearance less than 50 mL/min
* Corrected QT interval greater than 500 msec. on a 12-lead screening electrocardiogram

Observational Group (post-operative OIC screen/rescreen):

Exclude patients with:

* Fecal impaction
* Mechanical bowel obstruction
* Constipation not attributed to post-procedural opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute OIC in postoperative spinal surgery patients, specifically those undergoing 1-2 level anterior lumbar interbody fusion (ALIF) at Methodist Dallas Medical Center (MDMC)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Bowel Movement assessment | July 2021 - April 2022
  Percentage of patients with bowel movement (BM) within four hours of first RELISTOR dose or SOC bowel regimen
Post-treatment Bowel Movement | July 2021 - April 2022
  Time to Bowel Movement after first treatment

SECONDARY OUTCOMES:
Patient Assessment of Constipation Symptoms (PAC-SYM) | July 2021 - April 2022
  to measure patient's self-reported experience of symptoms and symptom severity in constipation pre-operatively and at patients post-operative follow-up
Treatment Satisfaction Questionnaire for Medication | July 2021 - April 2022
  to measure patients' satisfaction with medication
Bowel Function Diary | July 2021 - April 2022
  Daily Assessment Module: to measure constipation symptoms experienced in the past 24 hours during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Richard Meyrat, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Moody Brain and Spine Institute, Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No